CLINICAL TRIAL: NCT04690634
Title: The Changes of Body Fat Distribution in Obese Patients With Polycystic Ovary Syndrome After Laparoscopic Sleeve Gastrectomy
Brief Title: The Changes of Body Fat Distribution in Obese Patients With PCOS After LSG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai 10th People's Hospital (Other)
Responsible Party: Principal Investigator, Zhang Manna, Director, Principal Investigator, Clinical Professor, Shanghai 10th People's Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PCOS DEXA
Record Dates: First submitted 2020-12-20; First posted 2020-12-31 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2022-09

CONDITIONS: Polycystic Ovary Syndrome
Keywords: Laparoscopic Sleeve Gastrectomy; Body fat distribution; Dual-energy X-ray absorptiometry; Visceral adipose tissue
MeSH Terms: conditions — Polycystic Ovary Syndrome

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PCOS group (Experimental): obese female patients with Polycystic ovary syndrome. All participants underwent laparoscopic sleeve gastrectomy (LSG)
  Interventions: Procedure: laparoscopic sleeve gastrectomy (LSG)
- control group (Active Comparator): obese female patients without Polycystic ovary syndrome. All participants underwent laparoscopic sleeve gastrectomy (LSG)
  Interventions: Procedure: laparoscopic sleeve gastrectomy (LSG)

INTERVENTIONS:
Procedure: laparoscopic sleeve gastrectomy (LSG) — Multiple studies have indicated that laparoscopic sleeve gastrectomy (LSG) was superior to nonsurgical approaches for the treatment of obese PCOS patients over both the short and long term

SUMMARY:
Polycystic ovary syndrome (PCOS) is a common endocrine disorder, with a prevalence of 5% to 15% in premenopausal women. Patients with PCOS presents as abnormal menstruation, ovulation disorders and/or hyperandrogenemia, and often accompanied by insulin resistance and other metabolic abnormalities. Abdominal fat accumulation, overweightness and obesity are frequently present in patients with PCOS . Visceral adipose tissue (VAT) plays an important role in the pathogenesis of PCOS.Therefore，this study aim to investigate the changes of body fat distribution in obese women with PCOS after laparoscopic sleeve gastrectomy (LSG), and to explore the factors that may predict the changes in body fat distribution in PCOS patients after LSG.

DETAILED DESCRIPTION:
This study consecutively enrolled 153 patients with obesity aged 18-45 years (83 with PCOS and 70 control patients) who underwent LSG from May 2013 to September 2020 at the Department of Endocrinology, Shanghai Tenth People's Hospital, with a 12-month follow-up. Dual-energy X-ray absorptiometry (DEXA) was used to assess body fat distribution.

ELIGIBILITY:
Inclusion Criteria:

1. Fmale aged 18- 45;
2. Meet Rotterdam criteria(2003);
3. body mass index (BMI)≥30 kg/m2

Exclusion Criteria:

1. Gender is male;
2. Younger than 18 years old or older than 45 years old ;
3. secondary obesity due to endocrine disorders;
4. history of malignant tumors; 5）sever hepatic and renal disease;

6) concurrent participation in other clinical trials; 7) sever endocrine and hereditary diseases; 8) mental illnesses that rendered them unable to provide informed consent; 9) patients declining to undergo complete study testing.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 153 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
VAT mass | 12 months
  visceral adipose tissue (VAT) mass

SECONDARY OUTCOMES:
BMI | 12 months
  Body mass index (BMI) was calculated as follows: BMI = (body weight [kg])/(height [m2])
FBG | 12 months
  fasting blood-glucose in mmol/L
PBG | Baseline and 12 months
  postprandial blood-glucose in mmol/L
FINS | Baseline and 12 months
  fasting serum insulin in mU/L
PINS | Baseline and 12 months
  postprandial insulin in mU/L
ALT | Baseline and 12 months
  alanine aminotransferase in U/L
AST | Baseline and 12 months
  aspartate aminotransferase in U/L）
UA | Baseline and 12 months
  Uric acid in umol/L
CR | Baseline and 12 months
  Creatinine in umol/L
LDL-c | Baseline and 12 months
  low-density lipoprotein cholesterol in mmol/L
HDL-c | Baseline and 12 months
  high-density lipoprotein cholesterol in mmol/L
TC | Baseline and 12 months
  Total Cholesterol in mmol/L
TG | Baseline and 12 months
  Triglyceride in mmol/L
WHR | Baseline and 12 months
  waist-to-hip ratio (WHR) were calculated as follows: WHR = (waist circumference [cm]/(hip circumference [cm]).
HC | Baseline and 12 months
  Hip circumference
Ferriman-Gallwey score | Baseline and 12 months
  Ferriman-Gallwey score
Menstrual Cycles | Baseline and 12 months
  The number of menstrual cycles per year was defined as the number of menstruations during the last 12 months.
HOMA-IR | Baseline and 12 months
  homeostatic model assessment insulin resistance index
TT | Baseline and 12 months
  total testosterone in nmol/L
FT | Baseline and 12 months
  free testosterone (nmol/L)
DHEAS | Baseline and 12 months
  Dehydroepiandrosterone Sulfate (ug/dl)
SHBG | Baseline and 12 months
  sex hormone-binding globulin in nmol/L
FSH | Baseline and 12 months
  follicle-stimulating hormone in IU/L
LH | Baseline and 12 months
  luteinizing hormone in IU/L
WC | Baseline and 12 months
  waist circumference,

CONTACTS AND LOCATIONS:
Overall Officials: Shen Qu, Dr, Study Chair — Shang hai Tenth People's Hospital
Locations (1):
- Department of Endocrinology, Shanghai Tenth People's Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cai M, Gao J, Du L, Cheng X, Zhou D, Zhu J, Qu S, Zhang M. The Changes in Body Composition in Obese Patients with Polycystic Ovary Syndrome after Laparoscopic Sleeve Gastrectomy:a 12-Month Follow-up. Obes Surg. 2021 Sep;31(9):4055-4063. doi: 10.1007/s11695-021-05496-6. PMID 34152560
- See also: The Changes in Body Composition in Obese Patients with Polycystic Ovary Syndrome after Laparoscopic Sleeve Gastrectomy:a 12-Month Follow-up — https://pubmed.ncbi.nlm.nih.gov/34152560/